CLINICAL TRIAL: NCT02588872
Title: Hyaluronic Acid vs Platelet Rich Plasma: Prospective Double-blind Randomized Controlled Trial Comparing Clinical Outcomes and the Effects on Intra-articular Biology for the Treatment of Knee Osteoarthritis
Brief Title: Hyaluronic Acid vs Platelet Rich Plasma: Effects on Clinical Outcomes and Intra-articular Biology for the Treatment of Knee Osteoarthritis
Acronym: HA vs PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Cornell University (Other)
Responsible Party: Principal Investigator, Carla Edwards, Clinical Trials Investigator, Rush University Medical Center, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10012103-AM02
Record Dates: First submitted 2015-10-25; First posted 2015-10-28 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis, Knee
Keywords: platelet-rich plasma; hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronic Acid (HA) (Active Comparator): Hyaluronic acid administered as an intra-articular injection under ultrasound guidance as a series of three weekly injections to the affected knee. 3 weekly injections are of ultra high molecular weight hyaluronan (16mg) in a 2mL injection.
  Interventions: Biological: Hyaluronic Acid
- Platelet-rich Plasma (PRP) (Experimental): Platelet-rich plasma administered as an intra-articular injection under ultrasound guidance as a series of three weekly injections to the affected knee. 3 weekly injections are of leukocyte poor, buffer/additive free, singe spin, platelet-rich plasma averaging 4mL in volume.
  Interventions: Biological: Platelet-rich Plasma (PRP)

INTERVENTIONS:
Biological: Platelet-rich Plasma (PRP)
  Arms: Platelet-rich Plasma (PRP)
Biological: Hyaluronic Acid
  Arms: Hyaluronic Acid (HA)

SUMMARY:
In this, prospective, double-blind study, patients with mild to moderate symptomatic knee osteoarthritis will be randomized to receive either a series of leukocyte poor, platelet-rich plasma or hyaluronic acid injections under ultrasound guidance. Clinical data in the form of subjective outcome measures will be collected pre-treatment and at four time intervals across a 1-year period. Synovial fluid will also collected for analysis of pro- and anti-inflammatory markers pre-treatment, and at 12 and 24 weeks.

DETAILED DESCRIPTION:
The objective of this double-blind prospective randomized clinical trial is to compare the effects of PRP to HA in patients with mild to moderate OA using biologic and clinical correlates of outcomes associated with the treatment of OA. The investigators will test the null hypothesis that there are no differences in clinical outcomes as measured by validated clinical scoring systems for OA, nor is there any difference in intra-articular biology between groups of patients treated with HA and those treated with PRP over time.

This study was a prospective, randomized, double blind, comparative clinical trial with an allocation ratio of 1:1 that underwent IRB approval at the principal institution. Between 2011 and 2014 patients will be screened for participation. All comers with a diagnosis of osteoarthritis of the knee between 18 and 80 years of age will be screened.

Treatment and Evaluation Patients who meet inclusion criteria will be randomized via an electronic randomization process into two groups: one receiving intra-articular PRP and the other, intra-articular HA. Non-clinical staff will perform randomization, clinical staff performed the injections, and results and analyses will be performed by the primary research team. Patients and the primary research team performing analysis will be blinded to assignments. All patients will undergo a 10 ml blood draw for PRP preparation and a 3 ml peripheral blood draw for a complete blood count with leukocyte differential. This will be performed on patients who received HA to maintain patient blinding and to characterize the peripheral white blood cells (WBC) and platelet counts. A complete blood count (CBC) will be completed on PRP prior to injection to evaluate the fold increase in platelet concentration and to confirm rarity of red white blood cells. A synovial fluid aspirate of approximately 2cc will be performed under ultrasound guidance just prior to each PRP or HA injection for ELISA analysis of basal and post-treatment intra-articular environment. After treatment, patients will be instructed to limit the use of the leg for at least 24 hours and use cold therapy/icing for discomfort. During this treatment period rest or mild exertion activities (such as exercise bike, aquatic therapy) are recommended, followed by gradual return to sports or recreational activities as tolerated.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Mild to moderate unilateral, symptomatic osteoarthritis of the knee
* No recent (within 3 months) intra-articular intervention to the affected knee

Exclusion Criteria:

* Knee instability
* Varus/Valgus alignment >5 degrees
* Bilateral knee osteoarthritis
* Systemic inflammatory arthropathy
* Known history of anemia, coagulopathy, or present use of blood thinners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2011-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Cole BJ, Karas V, Hussey K, Pilz K, Fortier LA. Hyaluronic Acid Versus Platelet-Rich Plasma: A Prospective, Double-Blind Randomized Controlled Trial Comparing Clinical Outcomes and Effects on Intra-articular Biology for the Treatment of Knee Osteoarthritis. Am J Sports Med. 2017 Feb;45(2):339-346. doi: 10.1177/0363546516665809. Epub 2016 Oct 21. PMID 28146403

RESULTS

PARTICIPANT FLOW:
Groups:
- Hyaluronic Acid (HA): Hyaluronic acid administered as an intra-articular injection under ultrasound guidance as a series of three weekly injections to the affected knee. 3 weekly injections are of ultra high molecular weight hyaluronan (16mg) in a 2mL injection.
  Hyaluronic Acid
- Platelet-rich Plasma (PRP): Platelet-rich plasma administered as an intra-articular injection under ultrasound guidance as a series of three weekly injections to the affected knee. 3 weekly injections are of leukocyte poor, buffer/additive free, singe spin, platelet-rich plasma averaging 4mL in volume.
  Platelet-rich Plasma (PRP)
Period: Overall Study
Arm/Group | Hyaluronic Acid (HA) | Platelet-rich Plasma (PRP)
Started | 59 | 52
Completed | 59 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyaluronic Acid (HA) | Platelet-rich Plasma (PRP) | Total
Number analyzed (Participants) | 59 | 52 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.5) | 55.9 (10.4) | 56.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were a total of 12 patients that were lost to follow-up, 3 in the PRP group and 9 in the HA group thus the final numbers included in analysis was 99 total patients instead of 111.
  Participants
    number analyzed (Participants) | 50 | 49 | 99
    Female | 30 | 21 | 51
    Male | 20 | 28 | 48
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29 (6.4) | 27.4 (3.9) | 28.2 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: International Knee Documentation Committee Score (IKDC
Description: This is a scale from 1-100, 100 being high function and 1 being very poor function that will be assessed via paper questionnaire at the delineated time intervals. The Primary outcome assessed will be at an average of 1-year post treatment.
Time Frame: This will be assessed as a change from pre-treatment visit to 1 year post treatment.
Population: 9 HA patients and 3 PRP from the original cohort were lost to follow up which is why 50 HA and 49 PRP patients were included in final analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hyaluronic Acid (HA) | Platelet-rich Plasma (PRP)
Number analyzed (Participants) | 50 | 49
units on a scale | 65.5 (3.6) | 55.8 (3.8)

2. Secondary Outcome: Visual Analogue Scale (VAS)
Description: This is a scale from 1-100, 100 being the worst pain imaginable and 1 being no pain at all that will be assessed via paper questionnaire at the delineated time intervals. The Primary outcome assessed will be at an average of 1-year post treatment.
Time Frame: This will be assessed as a change from pre-treatment visit to 1 year post treatment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hyaluronic Acid (HA) | Platelet-rich Plasma (PRP)
Number analyzed (Participants) | 50 | 49
units on a scale | 57.3 (3.8) | 44 (4.6)

3. Secondary Outcome: Western Ontario and McMaster Universities Arthritis Index
Description: as for outcome 1
Time Frame: This will be assessed as a change from pre-treatment visit to 1 year post treatment. 6-weeks post-treatment, 6-months post treatment, and finally at 1-year post treatment will be documented for the purpose of trending data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hyaluronic Acid (HA) | Platelet-rich Plasma (PRP)
Number analyzed (Participants) | 50 | 49
units on a scale | 4 (0.6) | 3.02 (0.48)

4. Secondary Outcome: Lysholm Knee Score
Description: as for outcome 1
Time Frame: This will be assessed as a change from pre-treatment visit to 1 year post treatment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hyaluronic Acid (HA) | Platelet-rich Plasma (PRP)
Number analyzed (Participants) | 50 | 49
units on a scale | 55.8 (3.8) | 65.5 (3.6)

5. Secondary Outcome: Biologic Testing of Synovial Fluid Via ELISA Assays
Description: ELISA analysis will be performed for the following biological markers: IL-1β, IL-1ra, IL-6, IL-8, TNFα
Time Frame: Primary outcome will be change from pre-treatment to 6-month post treatment.
Population: IL-1B
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hyaluronic Acid (HA) | Platelet-rich Plasma (PRP)
Number analyzed (Participants) | 50 | 49
units on a scale | 0.14 (0.005) | 0.34 (0.16)

ADVERSE EVENTS:
Arm/Group | Hyaluronic Acid (HA) | Platelet-rich Plasma (PRP)
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/52
Other Adverse Events (participants affected / at risk) | 0/59 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No